CLINICAL TRIAL: NCT03368521
Title: The Benefit of Structured Triage of Patients in the Primary Health Care Seeking Care for Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: FoU Center Spenshult (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Low back pain_RCT_2017
Record Dates: First submitted 2017-11-14; First posted 2017-12-11 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Back pain screening group (Other): Includes the Group of patients where the care giver has used the back pain screening tests studied in order to judge how to proceed with rehabilitation, which level of rehabilitation is appropriate.
  Interventions: Other: Back pain screening test
- treatment as usual (No Intervention): The Group get treatment as usual, where the care giver base the rehabilitation plan without taking the scorings from the screening tool into consideration.

INTERVENTIONS:
Other: Back pain screening test — The care giver use the screening tool in order to score the back patient to three levels of risk. For each level of risk, one suggested type of care is provided; 1) simple advise; 2) physiotherapy; 3) multimodal rehabilitation. highest risk level includes multimodal intervention.
  Arms: Back pain screening group

SUMMARY:
This study aims to investigate if a low back pain screening tool is helpful for the caregivers to direct the rehabilitation in a more efficient way, at an earlier stage. Primary Health care centers in the municipality of Halmstad, Sweden will be enrolled to participate in the study as either "Control" or "intervention". The primary Health care centers who are enrolled taking part in the intervention, will use the provided screening tool when taking care of patients seeking care for low back pain. Scorings from the screening tool will "label" the patients as one of Three pre-defined risk levels. The caregiver will then use the provided risk level when deciding how to proceed the rehabilitation. Based on the risk level identified, the patient is directed to one of three levels of treatments - including simple advice; physiotherapy; or multimodal rehabilitation. The screening tool is used as a complement to the examination, allowing the physiotherapist /GP to decide how to proceed with rehabilitation using the back screening tool, together with Clinical examinations. The Control Group consists of patients recruited when seeking care for back pain at a Primary Health Care service who has been randomly selected as "Control". The care givers at the Control primary Health care will conduct as usual, not using the back pain screening tool in their Clinical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Seeking care for low back pain at any of the included primary Health care.

Exclusion Criteria:

* Red flags

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of physiotherapy treatments | 4 months after inclusion
  Number of treatments given by physiotherapist
Number of physiotherapy treatments | 12 months after inclusion
  Number of treatments given by physiotherapist

SECONDARY OUTCOMES:
back pain questionnaire - The Keele STarT Back Screening Tool | 4 months after inclusion
  The Keele STarT Back Screening Tool, is a prognostic tool helping clinicians identify risk factors for persistent back pain. 9 questions. Total score range from 0 to 9 (best- to worse)
back pain questionnaire - The Keele STarT Back Screening Tool | 12 months after inclusion
  The Keele STarT Back Screening Tool, is a prognostic tool helping clinicians identify risk factors for persistent back pain. 9 questions. Total score range from 0 to 9 (best- to worse)
back pain questionnaire - Pain distribution | 4 months after inclusion
  Pain distribution (numbers of marked regions and location) will be measured by a pain mannequin divided into 18 body regions.The patients mark each region with pain lasting more than three months during the past 12 months. The total number of regions giving a total score 0-18 (few to several regions, best- to worse).
back pain questionnaire - Pain distribution | 12 months after inclusion
  Pain distribution (numbers of marked regions and location) will be measured by a pain mannequin divided into 18 body regions.The patients mark each region with pain lasting more than three months during the past 12 months. The total number of regions giving a total score 0-18 (few to several regions, best- to worse).
back pain questionnaire - The Roland-Morris Disability Questionnaire | 4 months after inclusion
  The Roland-Morris Disability Questionnaire assess self-rated physical disability Total score range from 0-24 (best to worse disability)
back pain questionnaire - The Roland-Morris Disability Questionnaire | 12 months after inclusion
  The Roland-Morris Disability Questionnaire assess self-rated physical disability Total score range from 0-24 (best to worse disability)
work ability - Work productivity and activity impairment questionnaire (WPAI) | 4 months after inclusion
  Work productivity and activity impairment questionnaire (WPAI) with 6 questions assessing the impact of the disease on work and other daily activities during the previous 7 days (absenteeism, presenteeism, impaired activities outside work, and overall work impairment). Each component is expressed as percentage of impairment due to the disease (0-100%) where a higher percentage indicates a greater reduction.
work ability - Work productivity and activity impairment questionnaire (WPAI) | 12 months after inclusion
  Work productivity and activity impairment questionnaire (WPAI) with 6 questions assessing the impact of the disease on work and other daily activities during the previous 7 days (absenteeism, presenteeism, impaired activities outside work, and overall work impairment). Each component is expressed as percentage of impairment due to the disease (0-100%) where a higher percentage indicates a greater reduction.
work ability - The work ability index (WAI) | 4 months after inclusion
  The work ability index (WAI) single-item question concerned the item "current work ability compared with the lifetime best", with a possible score of 0 ("completely unable to work") to 10 ("work ability at its best")
work ability - The work ability index (WAI) | 12 months after inclusion
  The work ability index (WAI) single-item question concerned the item "current work ability compared with the lifetime best", with a possible score of 0 ("completely unable to work") to 10 ("work ability at its best")

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Bergman, PhD, Study Chair — FoU Center Spenshult
Locations (1):
- FoUSpenshult, Halmstad, Sweden